CLINICAL TRIAL: NCT03797001
Title: The Effects of Interleukin-1 Blockade On Exercise Capacity In Patients With Recently Decompensated Systolic Heart Failure
Brief Title: Interleukin-1 Blockade In Recently Decompensated Heart Failure - 2
Acronym: REDHART2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REDHART2 HM20014686
Record Dates: First submitted 2019-01-02; First posted 2019-01-08 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure, Systolic; Inflammation
Keywords: heart failure; inflammation; anakinra; exercise capacity
MeSH Terms: conditions — Heart Failure, Systolic; Inflammation; Heart Failure | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- anakinra (Experimental): Anakinra subcutaneous injection, 100 mg daily for 24 weeks
  Interventions: Drug: Anakinra
- placebo (Placebo Comparator): Placebo subcutaneous injection, daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra — 100 mg subcutaneous injection, daily for 24 weeks
  Arms: anakinra
Drug: Placebo — subcutaneous injection, daily for 24 weeks
  Arms: placebo

SUMMARY:
REDHART2 is a randomized, double-blinded, placebo-controlled trial to determine the effects of Anakinra on peak aerobic exercise capacity measured with a cardiopulmonary test after 24 weeks in patients with recently decompensated systolic heart failure and increased systemic inflammation.

DETAILED DESCRIPTION:
The REDHART2 (REcently Decompensated Heart failure Anakinra Response 2 Trial) study is a phase II clinical trial of anakinra or placebo to determine improvement in aerobic exercise capacity (by measuring maximal oxygen uptake (VO2)) in patients with recently decompensated systolic heart failure (HF). The recently completed pilot REDHART study showed anakinra treatment for 12 weeks led to a significant improvement in peak aerobic exercise capacity, whereas anakinra treatment for 2 weeks did not, and no significant changes were seen in placebo. The REDHART2 study is designed to expand and confirm the beneficial effect of sustained anakinra treatment (24 weeks) on peak VO2, and to explore the potential effect size on hospital readmissions for HF. The rationale of Interleukin-1 (IL-1) blockade with anakinra in heart failure stems from the evidence of a) reduced adverse cardiac remodeling and heart failure in animal models of acute myocardial infarction (AMI); b) reduced incidence of heart failure in patients with ST-segment elevation AMI; c) enhanced IL-1 activity in patients with heart failure, d) quenching of the acute inflammatory response in patients with acute decompensated heart failure, e) direct cardiodepressant effects of IL-1 in animal models, f) improved exercise capacity in pilot studies including patients with stable systolic heart failure, stable diastolic heart failure, and, recently decompensated systolic heart failure in the pilot REDHART study. Patients will be randomized 2:1 to active treatment, such that patients will be twice as likely to receive anakinra versus placebo.

ELIGIBILITY:
Inclusion Criteria:

All 6 criteria need to be met for enrollment of the patient in the study

1. Primary diagnosis for hospitalization is decompensated heart failure established as the finding at admission of both conditions listed below:

   * dyspnea or respiratory distress or tachypnea at rest or with minimal exertion;
   * evidence of elevated cardiac filling pressure or pulmonary congestion (at least one of the conditions must be met):
   * pulmonary congestion/edema at physical exam OR chest XRay;
   * plasma BNP levels ≥200 pg/mL;
   * invasive measurement of left ventricular end-diastolic pressure >18 mmHg or of pulmonary artery occluding pressure (wedge) >16 mmHg.
2. The patient has a prior documentation of impaired left ventricular systolic function (ejection fraction ≤40%) at most recent assessment by any imaging modality (within 12 months).
3. The patient is now clinically stable, euvolemic, and meets standard criteria for hospital discharge as documented by all the 3 conditions listed below:

   * absence of dyspnea or pulmonary congestion/distress at rest;
   * absence of pitting edema in the lower extremities, or in any other region;
   * stable hemodynamic parameters (blood pressure, heart rate).
4. The patient is of age ≥21 years old, and is willing and able to provide written informed consent.
5. The patient is willing and able to comply with the protocol (i.e., self-administration, or exercise test).
6. The patient has screening high sensitivity plasma C-reactive protein levels (hsCRP) >2 mg/L.

Exclusion Criteria:

Subjects will not be eligible if they meet any of the following 15 exclusion criteria.

1. The primary diagnosis for admission is NOT decompensated heart failure, including diagnosis of acute coronary syndromes, hypertensive urgency/emergency, tachy- or brady-arrhythmias.
2. Concomitant clinically significant comorbidities that would interfere with the execution or interpretation of the study including but not limited to acute coronary syndromes, uncontrolled hypertension or orthostatic hypotension, tachy- or brady-arrhythmias, acute or chronic pulmonary disease or neuromuscular disorders affecting respiration.
3. Recent (previous 3 months) or planned resynchronization therapy (CRT), or valve surgeries.
4. Previous or planned implantation of left ventricular assist devices or heart transplant.
5. Chronic use of intravenous inotropes.
6. Recent (<14 days) use of immunosuppressive or anti-inflammatory drugs (including oral corticosteroids at a dose of prednisone equivalent of 0.5 mg/kg/day but not including inhaled or low dose oral corticosteroids or non-steroidal anti-inflammatory drugs).
7. Chronic inflammatory disorder (including but not limited to rheumatoid arthritis, systemic lupus erythematosus).
8. Active infection (of any type), including chronic/recurrent infectious disease (i.e. HBV, HCV, and HIV/AIDS) - but excluding HCV+ with undetectable plasma RNA.
9. Active malignancy - excluding carcinoma in situ [any location] or localized non-melanoma skin cancer.
10. Any comorbidity limiting survival or ability to complete the study.
11. Stage V kidney disease or on renal-replacement therapy.
12. Neutropenia (<1,500/mm3 or <1,000/mm3 in African-American patients).
13. Pregnancy.
14. Angina, hypertension, arrhythmias, electrocardiograph (ECG) changes, or other non-cardiac limitations (i.e., peak respiratory exchange ratio VCO2/VO2 [RER]<1.0, reflecting sub-maximal test) that limit maximum exertion during CPX obtained during the baseline testing.
15. Hypersensitivity to Kineret or to E. coli derived products. 16) Evidence of COVID19 within the last 60 days or recent (21 days) exposure to close personal contact.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Van Tassell, PharmD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Derived] Van Tassell BW, Golino M, Canada JM, Markley R, Billingsley H, Del Buono M, Talasaz A, Thomas G, Chiabrando JG, Wohlford G, Dickson V, Kadariya D, Damonte JI, Ho AJ, Sedhai YR, Kontos E, Vecchie A, West JD, Corna G, Medina de Chazal H, Pinel S, Bressi E, Barron A, Dell M, Mbualungu J, Moroni F, Turlington J, Federmann E, Trankle C, Carbone S, Arena R, Abbate A. Resolution of Systemic Inflammation in Patients With Recently Decompensated Heart Failure With Reduced Ejection Fraction With and Without Interleukin-1 Blockade by Anakinra. Circ Heart Fail. 2025 Dec 23:e013546. doi: 10.1161/CIRCHEARTFAILURE.125.013546. Online ahead of print. PMID 41431894
- [Derived] Van Tassell B, Mihalick V, Thomas G, Marawan A, Talasaz AH, Lu J, Kang L, Ladd A, Damonte JI, Dixon DL, Markley R, Turlington J, Federmann E, Del Buono MG, Biondi-Zoccai G, Canada JM, Arena R, Abbate A. Rationale and design of interleukin-1 blockade in recently decompensated heart failure (REDHART2): a randomized, double blind, placebo controlled, single center, phase 2 study. J Transl Med. 2022 Jun 15;20(1):270. doi: 10.1186/s12967-022-03466-9. PMID 35706006
- [Derived] Sedhai YR, Patel NK, Mihalick V, Talasaz A, Thomas G, Denlinger BL, Damonte JI, Del Buono MG, Federmann E, Hardin M, Ibe I, Harmon M, Van Tassell B, Abbate A. Heart failure clinical trial enrollment at a rural satellite hospital. Contemp Clin Trials. 2022 Apr;115:106731. doi: 10.1016/j.cct.2022.106731. Epub 2022 Mar 11. PMID 35283262

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anakinra | Placebo
Started | 68 | 34
Completed | 57 | 27
Not Completed | 11 | 7
Not completed — Withdrawn due to COVID19 | 4 | 0
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anakinra | Placebo | Total
Number analyzed (Participants) | 68 | 34 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 23 | 74
  >=65 years | 17 | 11 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [47 to 65] | 58 [46 to 67] | 58 [47 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 26 | 66
  Male | 28 | 8 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 47 | 28 | 75
  White | 19 | 6 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 68 | 34 | 102

OUTCOME MEASURES:

1. Primary Outcome: Changes in Peak Oxygen Consumption (VO2)
Description: changes in peak oxygen consumption (VO2) after 24 weeks of treatment
Time Frame: baseline - 24 weeks
Population: patients with data available for primary outcome analysis
Measure: Median (Inter-Quartile Range); unit: mL/kg/min
Arm/Group | Anakinra | Placebo
Number analyzed (Participants) | 57 | 27
mL/kg/min | 1.50 [-0.15 to 3.35] | 1.20 [0.5 to 3.9]
Statistical Analysis 1: Comparison: Anakinra vs Placebo; Test type: Superiority; p = 0.60, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Anakinra | Placebo
All-Cause Mortality (participants affected / at risk) | 0/68 | 1/34
Serious Adverse Events (participants affected / at risk) | 12/68 | 6/34
Other Adverse Events (participants affected / at risk) | 11/68 | 7/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anakinra (N=68) | Placebo (N=34)
Death (Cardiac disorders) | 0 | 1
Heart failure hospitalization (Cardiac disorders) | 6 | 3
Any hospitalization (General disorders) | 12 | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anakinra (N=68) | Placebo (N=34)
Infection requiring antibiotic (Infections and infestations) | 11 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT03797001/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT03797001/ICF_001.pdf